CLINICAL TRIAL: NCT01603563
Title: Stepped Care for Young Children After Trauma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH092373-01A1 (NIH)
Record Dates: First submitted 2012-05-09; First posted 2012-05-23 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stepped Care; Trauma-Focused Cognitive Behavioral Therapy; Preschool children
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepped Care TF-CBT (Experimental): Patients will receive step one: 3 (1 hr.) in-office therapist-led sessions over 6 weeks, the parent-child workbook (Stepping Together), scheduled weekly phone meetings (15 minutes), and information from the National Child Traumatic Stress Network website (via web or paper for those without access). Children who do not meet responder status will receive step two: 9 (1 to 1.5 hr.) in-office therapist-directed sessions of TF-CBT over 6 to 8 weeks.
  Interventions: Behavioral: Stepped Care TF-CBT
- Standard TF-CBT (Active Comparator): Patients will receive 12 (1 to 1.5 hr.) standard weekly in-office therapist-directed sessions over 12 to 14 weeks (Phase II only). The 2 additional weeks allow for scheduling difficulty. Standard TF-CBT includes child, parent and conjoint parent-child sessions addressing the core trauma treatment components discussed in section a.3 (e.g. stress management, skill building, gradual exposure, & trauma narrative etc.).
  Interventions: Behavioral: Standard TF-CBT

INTERVENTIONS:
Behavioral: Stepped Care TF-CBT — Stepped Care TF-CBT patients will receive step one: 3 (1 hr.) in-office therapist-led sessions over 6 weeks, the parent-child workbook (Stepping Together), scheduled weekly phone meetings (15 minutes), and information from the National Child Traumatic Stress Network website (via web or paper for those without access). Children who do not meet responder status will receive step two: 9 (1 to 1.5 hr.) in-office therapist-directed sessions of TF-CBT over 6 to 8 weeks.
  Arms: Stepped Care TF-CBT
Behavioral: Standard TF-CBT — Standard TF-CBT patients will receive 12 (1 to 1.5 hr.) standard weekly in-office therapist-directed sessions over 12 to 14 weeks (Phase II only). The 2 additional weeks allow for scheduling difficulty. Standard TF-CBT includes child, parent and conjoint parent-child sessions addressing the core trauma treatment components discussed in section a.3 (e.g. stress management, skill building, gradual exposure, & trauma narrative etc.).
  Arms: Standard TF-CBT

SUMMARY:
The aim of this R34 study is to develop and test the feasibility of a Stepped Care intervention for young children with Posttraumatic Stress Disorder (PTSD). Phase I will focus on developing and testing the feasibility of Stepped Care Trauma-Focused Cognitive Behavioral Therapy (SC-TF-CBT) in a small open trial (N=10). Phase II will consist of a randomized controlled trial (N=54) examining the efficacy of SC-TF-CBT relative to standard Trauma-Focused Cognitive Behavioral Therapy (TF-CBT)on a number of outcome measures, treatment acceptability and satisfaction, and costs of treatment delivery. Findings from this pilot study will establish the feasibility and preliminary efficacy (see Kraemer et al., 2006) of SC-TF-CBT before progressing to a larger, randomized R01 to examine the effectiveness of SC-TF-CBT for early childhood PTSD.

DETAILED DESCRIPTION:
Young children who are exposed to traumatic events such as abuse, disasters, accidents, illnesses, injury and the death of a person close to them are at risk for developing PTSD. While effective treatments for childhood PTSD exist, novel interventions that are more accessible, efficient, and cost-effective are needed to improve access to evidence-based treatment. The purpose of this study is to develop and test the feasibility of an intervention called Stepped Care Trauma-Focused Cognitive Behavioral Therapy which has the potential to greatly improve service delivery approaches to make treatment more accessible and less costly, thereby reducing childhood PTSD and related societal impacts and costs.

ELIGIBILITY:
Inclusion Criteria:

1. Child must have experienced at least one traumatic event after the age of 36 months.
2. At least five Postttraumatic stress symptoms with one symptom of reexperiencing or one symptom of avoidance.
3. Child must be between 3 and 7 years of age at the time of enrollment.
4. The parent must be willing and able to participate in the treatment and complete informed consent.

Exclusion Criteria:

1. Psychosis, mental retardation, autism, or related pervasive developmental disorders in child or any condition that would limit the caregiver's ability to understand CBT and the child's ability to follow instructions.
2. Parent has had substance use disorder within the past 3 months.
3. Child or parent is suicidal (the DIPA will be used to screen for child suicidal ideation and the SCID-RV will be used to screen for parent suicide ideation; assessed by all available information). A delayed entry once the parent or child is stabilized (at least 6 months post suicidal) and not having suicidal ideation will be allowed.
4. Child or parent is not fluent in English.
5. Child is currently taking psychotropic medication and is not on a stable medication regimen for at least 4 weeks prior to admission to the study. If appropriate, a delayed entry will be allowed so that once a child is on a stable dosage the child may be enrolled in the study.
6. Child is receiving trauma-focused psychotherapy when study treatment is provided.
7. Parent or caregiver who would be treatment participant was the perpetrator, or the child was perpetrated by a person who still lives in the home (e.g. mother's boyfriend, sibling).

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Posttraumatic stress symptoms | baseline, week 14, and 3 month follow up
  Change from baseline in Diagnostic Preschool Infant Assessment PTSD module (DIPA; Scheeringa, 2010) and in the Trauma Symptom Checklist for Young Children (Briere et al., 2001) at 14 weeks and 3 month follow up

SECONDARY OUTCOMES:
Externalizing behaviors | baseline and week 14 and 3 month follow up
  Change from baseline in the Child Behavior Checklist (Achenbach & Rescorla, 2000) externalizing behaviors at 14 weeks and 3 month follow up
Internalizing behaviors | baseline, week 14 and 3 month follow up
  Change from baseline in the Child Behavior Checklist (Achenbach & Rescorla, 2000) internalizing behaviors at week 14 and 3 month follow up
Independent Evaluator-rated PTSD symptom and impairment severity | baseline, week 14 and 3 month follow up
  Change from baseline in clinical global impression severity (NIMH, 1985)at week 14 and 3 month follow up
Global improvement | baseline, week 14 and 3 month follow up
  Change from baseline in clinical global impression - improvement (Guy, 1976)at week 14 and 3 month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Alison A Salloum, PhD, Principal Investigator — University of South Florida
Locations (1):
- Crisis Center of Tampa Bay, Tampa, Florida, United States

REFERENCES:
- [Derived] Salloum A, Wang W, Robst J, Murphy TK, Scheeringa MS, Cohen JA, Storch EA. Stepped care versus standard trauma-focused cognitive behavioral therapy for young children. J Child Psychol Psychiatry. 2016 May;57(5):614-22. doi: 10.1111/jcpp.12471. Epub 2015 Oct 7. PMID 26443493